CLINICAL TRIAL: NCT01489748
Title: An Open-Label, Observational, Multicenter Study to Evaluate the Impact of AVONEX PEN Autoinjector Therapy on Work Capacity of Multiple Sclerosis Patients in Canada
Brief Title: Canadian Avonex PEN Productivity Study
Acronym: CAPPS
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: CAN-AVX-11-10239
Record Dates: First submitted 2011-12-01; First posted 2011-12-12 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is primarily designed to evaluate the impact of AVONEX PEN autoinjector on work capacity of participants with multiple sclerosis (MS) starting on this device. This study will also evaluate as secondary endpoints various patient-reported outcomes over the short-term (1 month), including adherence, treatment satisfaction and convenience, and the long-term (12 and 24 months), including adherence, persistence, quality of life (QOL), treatment satisfaction and convenience. It will also assess health resource utilization by MS participants starting on AVONEX PEN autoinjector, as well as overall safety/tolerability, and will correlate all secondary outcomes with the primary (i.e., work capacity).

ELIGIBILITY:
Key Inclusion Criteria:

* Must be prescribed AVONEX PEN as per local labeling (Product Monograph) and enrolled in MS Alliance (MSA) program
* If being switched from another DMT, must be on this DMT for at least 6 months
* Last DMT the subject is switched from must be injectable
* Must be able to physically demonstrate use of the AVONEX PEN autoinjector device and be able to self-administer the injections
* Must give written informed consent. If required by local law, candidates must also authorize the release and use of protected health information (PHI)
* Must be able to understand and comply with the protocol

Key Exclusion Criteria:

* Female subjects considering becoming pregnant while in the study or who are currently pregnant or breast-feeding
* Current enrollment in any investigational study involving drug, biologic or non-drug therapy
* Participation in other clinical studies within the past 6 months
* Treatment with immunosuppressive regimens (e.g. cyclophosphamide, azathioprine, methotrexate or mitoxantrone) or with intravenous immunoglobulin (IVIg) in the last 6 months
* The most recent DMT the subject is switched from is non-injectable (i.e., oral)
* Other unspecified reasons that, in the opinion of the Investigator or Sponsor, make the subject unsuitable for enrollment

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Enrollment will consist of approximately 500 participants who have been prescribed AVONEX PEN in accord with its labeling (Product Monograph). This will include participants who are naïve to disease modifying therapies (DMTs) as well as those who are being switched from another injectable DMT.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in work capacity | 2 years
  Work capacity will be assessed by a telephone-based survey which consists of 10 questions asking participant's about the effect of MS on their ability to work and perform regular activities.

SECONDARY OUTCOMES:
Number of participants with hospital and emergency episodes of care | -1 year, 1 year
Number of missed injections | 1 month, 1 year, 2 years
Number of participants who discontinued treatment | 1 year, 2 years
Change from Baseline in Global Quality of life score | 1 year, 2 years
  Quality of life will be assessed by a Multiple Sclerosis Quality of Life (MSQOL) questionnaire. This 54-item questionnaire addresses overall health and daily activities.
Change from Baseline in participants' satisfaction with the device | 1 month, 1 year, 2 years
  Participant satisfaction will be measured using a 10-item satisfaction questionnaire.
Change from Baseline in ease of use of the device | 1 month, 1 year, 2 years
  Ease of use will be assessed on a scale from 0 (extremely difficult) to 10 (extremely easy).
Number of participants with injection site reactions (ISRs) | 1 month, 1 year, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Central Contact, Burlington, Ontario, Canada